CLINICAL TRIAL: NCT02241811
Title: Deep Diabetic Foot Wound Treatment With Hydrogel Including 3% Sodium Pentaborate Pentahydrate
Brief Title: Wound Treatment With 3% Sodium Pentaborate Pentahydrate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Erhan Aysan, MD Prof., SB Istanbul Education and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Boron wound
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2018-09

CONDITIONS: Wound Healing
Keywords: Diabetic; Foot; Wound; Sodium pentaborate pentahydrate; Hydrogel
MeSH Terms: conditions — Wounds and Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): After wound dressing we applied hydrogel without any active ingredient everyday for two months. The same doctor observed and took photo of the wounds every week in the outpatients clinic.
  Interventions: Drug: Placebo
- 3% Sodium Pentaborate Pentahydrate (Experimental): For the interventional group after wound dressing we applied hydrogel with 3% Sodium pentaborate pentahydrate everyday for two months. The same doctor observed and took photo of the wounds every week in the outpatients clinic.
  Interventions: Drug: 3% Sodium Pentaborate Pentahydrate

INTERVENTIONS:
Drug: 3% Sodium Pentaborate Pentahydrate — For the interventional group after wound dressing we applied hydrogel with 3% Sodium pentaborate pentahydrate everyday for two months. The same doctor observed and took photo of the wounds every week in the outpatients clinic.
  Other Names: 3% Sodium Pentaborate Pentahydrate group, Control Group
  Arms: 3% Sodium Pentaborate Pentahydrate
Drug: Placebo — Hydrogel without 3% Sodium Pentaborate Pentahydrate
  Arms: Control

SUMMARY:
Chronic foot wounds which is very difficult to treat are common especially in diabetic and peripheral arterial or venous insufficiency patients. This research is aim to observe the foot wound's recovery with 3% Sodium pentaborate pentahydrate hydrogel.

DETAILED DESCRIPTION:
Chronic foot wounds which is very difficult to treat are common especially in diabetic and peripheral arterial or venous insufficiency patients. For these reason we prepared a hydrogel formulations.

Gel preparation:

Hydrogel formulations were prepared by dispersing 1%(w/v) carbopol polymer (Carbopol Ultrez-21, Lubrizol, USA) in distilled water. Neutralization buffer (1.6g of 1M sodium hydroxide solution for 1L polymer-water suspension) was used for the gelation of the polymer. Sodium pentaborate pentahydrate (3% w/v), F68 (2% w/v) and F127 (2% w/v) were mixed into the blank hydrogel and stored at 4 °C until it completely dissolved (approximately 24 h). pH of the hydrogel formulation was set to 6.5-7.0 using 1M sodium hydroxide. The hydrogel without any active ingredient was used as negative control (vehicle).

For the first group after wound dressing we applied hydrogel with 3% Sodium pentaborate pentahydrate, and for the control group after wound dressing we applied hydrogel without any active ingredient everyday for two months. The same doctor observed and took photo of the wounds every week in the outpatients clinic.

ELIGIBILITY:
Inclusion Criteria:

Diabetic Foot wounds

Exclusion Criteria:

Child

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Wound healing, Complication | 2 months
  observation of wound healing and complications

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Aysan, MD Prof., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)